CLINICAL TRIAL: NCT02965482
Title: Volumetric Versus Standard Two Minute Tidal Breathing Methodology for Methacholine Challenge Testing
Brief Title: Investigation of Novel Procedure for Methacholine Challenge Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, MD, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MCT-SOLOWRIGHT-13
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: methacholine, airway hyperresponsiveness
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerogen Solo (Active Comparator): Volumetric method of methacholine challenge testing performed using the Aerogen Solo nebulizer
  Interventions: Device: Aerogen Solo Nebulizer
- Wright (Active Comparator): Two-minute tidal breathing method of methacholine challenge testing performed using the Wright nebulizer
  Interventions: Device: Wright Nebulizer

INTERVENTIONS:
Device: Wright Nebulizer — Roxon Medi-Tech, Montreal, QC, Canada
  Arms: Wright
Device: Aerogen Solo Nebulizer — Aerogen Ltd., Galway, Ireland
  Arms: Aerogen Solo

SUMMARY:
The study will compare a novel volumetric method (performed with the Aerogen Solo vibrating mesh nebulizer) with the standard two-minute tidal breathing protocol (performed with the Wright jet nebulizer) for methacholine challenge testing. The results will then give an indication as to whether the novel technique accurately assesses a given dose of methacholine with the new Aerogen Solo device. In addition, the reproducibility of test results with each method will be examined. Altogether, the findings from this investigation may provide means for better standardization of current testing guidelines.

DETAILED DESCRIPTION:
Fifteen asthmatics will be recruited and tested at the University of Saskatchewan for this randomized, two-way crossover study. Two testing methodologies will be performed, the volumetric method with the Aerogen Solo nebulizer and the two-minute tidal breathing method with the Wright nebulizer.

Participants will undergo four methacholine challenges plus a screening methacholine challenge. However, screening is omitted with participants who have completed a methacholine challenge in the last six months. Of the four study challenges, two will utilize the Wright nebulizer with the two-minute tidal breathing method outlined in the 1999 American Thoracic Society Guidelines for Methacholine Challenge Testing. The remaining two challenges will utilize the Aerogen Solo nebulizer with the volumetric method. The timing of the spirometric manoeuvers and the duration of each inhalation cycle will be consistent with both testing methods. Each challenge will be stopped when the participant's forced expiratory volume in 1 second (FEV1) drops by at least 20%. This allows determination of aPC20 (provocative concentration of methacholine causing a 20% fall in FEV1), which will be converted to aPD20 (provocative dose). A minimum 24-hour washout period between challenges will be used.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older
* Stable asthma
* Baseline methacholine PC20 less than or equal to 16mg/mL
* Baseline lung function equal or greater than 65% of predicted FEV1

Exclusion Criteria:

* Use of long-acting bronchodilators within 7 days of visit 1
* Pregnant or nursing women
* Cardiovascular problems
* Upper respiratory tract infection within 4 weeks of visit 1
* Allergy-induced asthma exacerbation within 4 weeks of visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Methacholine PD20 values of two nebulizers, each with a different testing protocol | 2 weeks
  Do the nebulizers produce similar responses at the same dose

SECONDARY OUTCOMES:
Comparability of PD20 values with a single nebulizer over two methacholine challenges | 2 weeks
  Does a nebulizer produce similar PD20 results with repeat testing

CONTACTS AND LOCATIONS:
Overall Officials: Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Asthma Research Lab - University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No